CLINICAL TRIAL: NCT06843408
Title: A Phase 1b/2, Open-Label, Multicenter Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Axatilimab Monotherapy in Chinese Participants With Recurrent or Refractory Active Chronic Graft-Versus-Host Disease After Systemic Therapy
Brief Title: A Ph1b/2 Study of Axatilimab Monotherapy in Chinese Participants With Recurrent or Refractory cGVHD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA34176-204
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1 Safety Evaluation (Experimental): Axatilimab at the protocol-defined dose.
  Interventions: Drug: INCA034176
- Part 2 Efficacy Evaluation (Experimental): Axatilimab at the protocol-defined dose.
  Interventions: Drug: INCA034176

INTERVENTIONS:
Drug: INCA034176 — IV infusion
  Other Names: Axatilimab

SUMMARY:
This study will be conducted to evaluate the safety, efficacy, and pharmacokinetics of axatilimab monotherapy in Chinese participants with recurrent or refractory active chronic graft-versus-host disease after systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age at the time of signing the ICF.
* Ability to comprehend and willingness to sign a written ICF for the study.

  • For participants 12 to 17 years old: A parent/guardian must provide consent for pediatric participants; when applicable, pediatric participants should also sign an assent form.
* Chinese participants who are allo-HSCT recipients with active, refractory, or recurrent cGVHD requiring systemic immune suppression despite prior systemic therapy, including corticosteroids and at least 1 other appropriate treatment for refractory or recurrent cGVHD.

  * Active cGVHD is defined as the presence of signs and symptoms of cGVHD per the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD (Jagasia et al 2015).
  * Refractory disease is defined as meeting any of the following criteria:

    * The development of 1 or more new sites of disease while being treated for cGVHD.
    * Progression of existing sites of disease despite at least 1 month of standard or investigational therapy for cGVHD.
    * Participants who did not achieve a response within 3 months on prior therapy for cGVHD and for whom the treating physician believes a new systemic therapy is required.
  * Recurrent cGVHD is defined as active, symptomatic disease (after an initial response to prior therapy) based on the NIH 2014 consensus criteria (Lee et al 2015) by organ-specific or global assessment or for which the physician believes a new line of systemic therapy is required.
* Participants may have persistent, active aGVHD and cGVHD manifestations (overlap syndrome), as defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.
* Karnofsky performance score of ≥ 60 (if aged 16 years or older); Lansky performance score of ≥ 60 (if aged younger than 16 years).
* Adequate organ and bone marrow functions evaluated during the 14 days prior to the start of study treatment as follows:

  * Absolute neutrophil count ≥ 1.0 × 109/L (without growth factors within 1 week of study entry).
  * Platelet count ≥ 50 × 109/L (without growth factor or transfusion within 2 weeks of study entry).
  * ALT and AST ≤ 2.5 × ULN and total bilirubin ≤ 1.5 × ULN. Note: For participants with suspected or documented liver cGVHD: ALT and AST ≤ 5 × ULN and total bilirubin ≤ 1.5 × ULN.
* Creatinine clearance ≥ 30 mL/min/1.73 m2 based on the Cockcroft-Gault formula in adult participants and the Schwartz formula in pediatric participants.
* Concomitant use of a systemic corticosteroid is allowed but not required. Topical and inhaled corticosteroid agents are allowed. If a participant is taking a corticosteroid, it must be a stable dose for at least 2 weeks prior to the start of study treatment.
* Concomitant use of CNIs or mTOR inhibitors is allowed but not required (the inhibitor may have been started either for prophylaxis or for treatment of cGVHD; the reason for initiating treatment must be recorded in the database). If a participant is taking a CNI or an mTOR inhibitor, the following criteria must be met:

  * Must be a stable dose for at least 2 weeks prior to the start of study treatment.
  * The dose must be within the therapeutic range.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

  * Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children from screening through 90 days (a spermatogenesis cycle) after the last dose of study treatment and must refrain from donating sperm during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants who are WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test before the first dose on Day 1 and must agree to take appropriate precautions to avoid pregnancy from screening through 30 days (1 menstrual cycle) after the last dose of study treatment and must refrain from donating oocytes during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants not considered to be of childbearing potential as defined in the protocol are eligible.

Exclusion Criteria:

* Has aGVHD without manifestations of cGVHD.
* Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
* History of acute or chronic pancreatitis.
* Active symptomatic myositis.
* History or other evidence of severe illness, uncontrolled infection, allergy to excipients (see formulation details in the IB), or any other conditions that would make the participant, in the opinion of the investigator, unsuitable for the study.
* Positive HIV status.
* History of latent or active TB, including either one of following:

  * Signs or symptoms suggestive of active TB upon medical history and/or physical examination.
  * Recent close contact with a person with active TB.
* Positive QuantiFERON and/or T-spot TB test at screening.
* Active HBV or HCV infection that requires treatment, or at risk for HBV reactivation (ie, positive HBsAg). Participants with negative HBsAg and positive total HBcAb and/or HBsAb should be excluded if quantitative HBV DNA test result is ≥ 20 IU/mL at the time of screening. Participants who are positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years before Cycle 1 Day 1 unless previously treated with curative intent (eg, completely resected basal cell or squamous cell carcinoma of the skin, resected in situ cervical malignancy, resected breast ductal carcinoma in situ, or low-risk prostate cancer after curative resection) and approved by the sponsor's medical monitor.
* Pregnant or breastfeeding.
* Previous exposure to CSF-1R targeted therapies.
* Use of any agent other than corticosteroids, CNIs, or mTOR inhibitors for the treatment of cGVHD within 2 weeks or 5 half-lives, whichever is shorter, prior to the start of study treatment.
* Has received an investigational treatment within 28 days prior to the start of study treatment.
* Currently participating in any other interventional study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event, occurring after the first dose.
Objective Response in the First 6 Cycles | Up to Cycle 7 (Day 169)
  The overall response rate will be assessed by the number of participants with objective response by Cycle 7 (28-day cycles), Day 1, with responses defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.

SECONDARY OUTCOMES:
Proportion of participants with a ≥ 7-point improvement in modified Lee symptom scale (mLSS) score | Up to 2 years
Overall Response Rate | Up to 2 years
  Defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.
Duration of Response | Up to 2 years
  Defined as the time from initial response of partial response or complete response until documented progression of cGVHD, start of new therapy, or death due to any cause, whichever occurs first.
Organ-specific Response Rate | Up to 2 years
  Organ-specific response is defined as the number of participants with objective response for the nine individual organs based on 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD (skin, eyes, mouth, esophagus, upper gastrointestinal [GI], lower GI, liver, lungs and joints and fascia).
Percent reduction in average daily dose (or equivalent) of corticosteroids | Up to 2 years
Proportion of participants who discontinue corticosteroid use | Up to 2 years
Percent reduction in average daily dose (or equivalent) of calcineurin inhibitors | Up to 2 years
Discontinuation of calcineurin inhibitor use after study entry. | Up to 2 years
Axatilimab pharmacokinetic (PK) in Plasma | Up to 2 years and 30 days
  Axatilimab concentration in plasma.
Change from baseline in colony-stimulating factor-1 (CSF-1) and interleukin (IL)-34 levels and its association with cGVHD response. | Up to 2 years
Change from baseline in circulating monocyte number and phenotype (CD14/16). | Up to 2 years
Number of Participants with Anti-Drug Antibody (ADA) | Up to 2 years and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (9):
- China (9):
  - Peking University People'S Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - The Second Affiliated Hospital, Army Medical University (Xinqiao Hospital), Chongoing
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Shanghai Children'S Medical Center, Shanghai
  - Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Ph1b/2 Study of Axatilimab Monotherapy in Chinese Participants With Recurrent or Refractory cGVHD — https://incyteclinicaltrials.com/studies/inca34176-204